CLINICAL TRIAL: NCT07249450
Title: Comparison of Sonic and Ultrasonic Activation of Irrigation Solutions on the Healing of Teeth With Apical Periodontitis
Brief Title: Comparison of Sonic and Ultrasonic Activation on Healing of Apical Periodontitis
Acronym: SONIC-ULTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Çuhadar Beşiroğlu (Other)
Responsible Party: Sponsor-Investigator, Hilal Çuhadar Beşiroğlu, DDS, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/164
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Apical Periodontitis
Keywords: Apical Periodontitis; Periapical Healing; Sonic Activation; Passive Ultrasonic Activation
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: Prospective
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sonic Activation (Experimental): Sonic irrigation activation using Micron TA-200 with EDDY tips
  Interventions: Procedure: Sonic Activation Irrigation
- Ultrasonic Activation (PUI) (Experimental): Passive ultrasonic irrigation using Ultra X activator
  Interventions: Procedure: Passive Ultrasonic Irrigation (PUI)
- Conventional Needle Irrigation (Control) (Active Comparator): Manual syringe irrigation using a 30-gauge side-vented needle
  Interventions: Procedure: Conventional Needle Irrigation

INTERVENTIONS:
Procedure: Sonic Activation Irrigation — Root canal irrigation activated sonically using EDDY tips (25/.04, VDW GmbH, Munich, Germany) attached to the Micron TA-200 sonic device. The tip was positioned 2 mm short of the WL. Sodium hypochlorite (2.5%), EDTA (17%), and chlorhexidine (2%) solutions were sequentially activated according to the study protocol.
  Arms: Sonic Activation
Procedure: Passive Ultrasonic Irrigation (PUI) — Irrigation activation performed with an ultrasonic activator (Ultra X, Eighteeth, China) using 21 mm silver tips with 2% taper. The tip was positioned 2 mm short of the WL. Sodium hypochlorite (2.5%), EDTA (17%), and chlorhexidine (2%) were activated sequentially following the standardized protocol.
  Arms: Ultrasonic Activation (PUI)
Procedure: Conventional Needle Irrigation — Manual syringe irrigation performed using a 30-gauge side-vented needle inserted 1 mm short of the WL. The canals were irrigated sequentially with sodium hypochlorite (2.5%), EDTA (17%), and chlorhexidine (2%) without any activation.
  Arms: Conventional Needle Irrigation (Control)

SUMMARY:
The goal of this clinical trial is to learn whether two different irrigation activation methods - passive ultrasonic irrigation (PUI) and sonic activation - help periapical healing in root canal treatments of single-rooted teeth with apical periodontitis.

Researchers will also compare these methods with the traditional needle irrigation technique.

The main questions this study aims to answer are

Do sonic irrigation activation or PUI activation methods lead to faster or better early periapical healing compared with traditional needle irrigation?

Is there any difference in healing volume measured by cone-beam computed tomography (CBCT) after 6 months?

Participants in this study will:

Adults with single-rooted teeth showing apical periodontitis (PAI ≥ 3),

Receive root canal treatment using either PUI, sonic activation, or traditional needle irrigation (assigned randomly).

Participants will have CBCT scans before treatment and again at 6 months to measure changes in lesion volume.

Researchers will analyze the 3D images using specialized software to calculate periapical lesion volumes before and after treatment. The study will evaluate how much the lesion size decreases in each group and whether any activation method improves healing compared with standard irrigation.

DETAILED DESCRIPTION:
Apical periodontitis (AP) develops as a consequence of pulpal infection and the subsequent host inflammatory response. The success of root canal treatment depends greatly on eliminating intraradicular biofilm and preventing reinfection. Adjunctive activation of irrigants-such as sonic or passive ultrasonic irrigation-has been proposed to enhance irrigant penetration, debris removal, and overall microbial disruption compared with conventional needle irrigation. This randomized, three-armed, parallel clinical trial evaluates whether sonic or ultrasonic activation of irrigating solutions leads to superior early periapical healing in single-rooted teeth diagnosed with AP. The study is based on the biological premise that activation improves irrigant replacement dynamics, acoustic streaming, and penetration into anatomically complex spaces that standard needle irrigation may not adequately reach. All participants received standardized root canal treatment using contemporary instrumentation, irrigation solutions, and obturation materials. The three intervention groups differed only in the method used to activate irrigants during the final cleaning phase. This uniformity ensured that any differences in healing outcomes reflect the effect of activation rather than variations in clinical technique. Early healing was assessed volumetrically using cone-beam computed tomography (CBCT), which enables three-dimensional visualization of periapical tissues and provides a sensitive measure of lesion change over time. Volumetric analysis was performed with a predefined workflow to ensure reproducibility, including blinded assessment to minimize bias. The study focuses on quantifying the reduction in periapical lesion volume at 6 months and exploring whether sonic or ultrasonic activation offers measurable advantages in early tissue healing compared with conventional irrigation. The findings aim to contribute to evidence-based endodontic protocols, particularly regarding the role of adjunctive activation techniques in improving periapical healing following root canal treatment.

ELIGIBILITY:
Inclusion Criteria:• American Society of Anesthesiologists physical status classification system (ASA) class I and II

* Individuals between 13 and 65 years of age
* Good oral hygiene

Tooth-related:

* Single-rooted teeth
* Sufficient amount of coronal tooth structure
* Probing depth of ≤ 4 mm
* Presence of Apical periodontitis (AP) on radiographs
* Asymptomatic teeth
* Periapical Index (PAI) score ≥ 3
* Negative response to pulp vitality tests
* Mature teeth

Exclusion Criteria:• ASA class III or higher

* Pregnancy or lactation
* Individuals with mental retardation
* Allergy to Sodium hypochlorite (NaOCl), Chlorhexidine (CHX), or latex

Tooth-related:

* Extensive structural loss that cannot be restored with a filling
* Presence of subgingival caries
* Teeth previously treated with root canal therapy
* Fractured or cracked teeth due to trauma
* Non-vital teeth without radiographic evidence of AP
* Immature teeth
* Positive response to pulp vitality tests
* Presence of internal or external root resorption detected on radiographs
* Increased mobility due to insufficient bone support

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Title: Change in Apical Lesion Volume Measured by Cone-Beam Computed Tomography (CBCT) | Baseline to 6 months post-treatment
  Volumetric change of apical periodontitis (AP) lesions in single-rooted teeth between baseline (pre-treatment) and 6-month follow-up, measured using 3D Doctor software on CBCT scans (Morita 3D Accuitomo 170). The measurement unit is cubic millimeters (mm³).
  Outcome Type: Continuous (quantitative)
  Statistical Method: Wilcoxon signed-rank test for within-group comparison; Kruskal-Wallis test for between-group analysis.

SECONDARY OUTCOMES:
Percentage Reduction in Apical Lesion Volume | Baseline to 6 months post-treatment
  Percent change (%) in lesion volume between baseline and 6-month follow-up, representing the proportion of lesion reduction relative to the initial volume. Healing is classified as complete (100%), partial (>25%), or uncertain (<25%) based on CBCT volumetric analysis.
Radiographic Healing Status | 6 months post-treatment
  Qualitative classification of periapical healing on CBCT and digital periapical radiographs into:
  1. complete healing (normal periodontal ligament space),
  2. partial healing (volume reduction),
  3. uncertain healing (<25% reduction),
  4. no healing or increased lesion size.

OTHER OUTCOMES:
Adverse Events During and After Treatment | Throughout treatment and follow-up period (baseline to 6 months)
  Number and type of clinical complications during or after endodontic treatment (flare-ups, swelling, restoration loss, or tooth fracture).

CONTACTS AND LOCATIONS:
Overall Officials: Işıl Kaya Büyükbayram, DDS, PhD, Study Director — Istanbul Aydın University, Faculty of Dentistry, Department of Endodontics; Hilal Cuhadar Besiroglu, DDS, Principal Investigator — Istanbul Aydın University, Faculty of Dentistry Department of Endodontics
Locations (1):
- Istanbul Aydın University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogan MU, Aricioglu B, Kose TE, Cikman AS, Oksuzer MC. Association between the irrigation-agitation techniques and Periapical Healing of large periapical lesions: a Randomized Controlled Trial. Clin Oral Investig. 2024 Jun 15;28(7):376. doi: 10.1007/s00784-024-05758-4. PMID 38878107
- [Background] Arikan NS, Hepsenoglu YE, Ersahan S, Ozcelik F. Periradicular repair after single-visit root canal treatment using sonic irrigant activation of teeth with apical periodontitis. Clin Oral Investig. 2024 Nov 26;28(12):656. doi: 10.1007/s00784-024-06059-6. PMID 39589537
- See also: Association between the irrigation-agitation techniques and Periapical Healing of large periapical lesions: a Randomized Controlled Trial — https://doi.org/10.1007/s00784-024-05758-4